CLINICAL TRIAL: NCT02077530
Title: Metabolic Syndrome Cohort in Korea
Status: Withdrawn | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Associate Professor, Korea University Anam Hospital
Other Study IDs: MS in KUMC
Record Dates: First submitted 2014-03-02; First posted 2014-03-04 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Metabolic Syndrome
Keywords: Patients with metabolic syndrome age between 30 to 64: Central obesity (Men ≥ 90 cm Women ≥ 85 cm), Plasma triglycerides ≥ 150 mg/dL; HDL cholesterol Men < 40 mg/dL, Women < 50 mg/dL, Blood pressure ≥130/85 mm Hg (or treatment for hypertension),; Fasting plasma glucose ≥ 100 mg/dL
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

SUMMARY:
Patients with metabolic syndrome living in Seoul area are included in this prospective registry for more than 10 years. All enrolled patients undergo thorough medical history survey. Enrolled patients will have coronary CT, 2D echocardiogram, treadmill test, pulse wave velocity, augmentation index, carotid intima-media thickness, and abdominal fat mass evaluation. Moreover, lipid profiles and inflammatory markers such as hsCRP, IL-6, TNF-alpha, VCAM-1, ICAM-1, adiponectin, MMP-9 will be measured. All participants will repeat the test and survey every year in Korea University Hospital.

ELIGIBILITY:
Inclusion Criteria: 3 out of 5 criteria

* Central obesity: Men ≥ 90 cm Women ≥ 85 cm
* Plasma triglycerides ≥ 150 mg/dL
* HDL cholesterol Men < 40 mg/dL, Women < 50 mg/dL
* Blood pressure ≥130/85 mm Hg (or treatment for hypertension)
* Fasting plasma glucose ≥ 100 mg/dL
* Age between 30 to 64
* Consent to our registry protocol

Exclusion Criteria:

* Patients who could not undergo coronary CT, 2D echocardiogram, treadmill test, and pulse wave velocity.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with metabolic syndrome living in Seoul area
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 10 years
  Cardiovascular events such as fatal and non-fatal myocardial infarction, heart failure, need for coronary and peripheral revascularization, stroke, all-cause death, and cardiac death.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital Metabolic Syndrome Research Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho DH, Kim MN, Joo HJ, Shim WJ, Lim DS, Park SM. Visceral obesity, but not central obesity, is associated with cardiac remodeling in subjects with suspected metabolic syndrome. Nutr Metab Cardiovasc Dis. 2019 Apr;29(4):360-366. doi: 10.1016/j.numecd.2019.01.007. Epub 2019 Jan 29. PMID 30782509
- [Derived] Lee D, Joo HJ, Jung HW, Lim DS. Investigating potential mediator between statin and coronary artery calcification. PLoS One. 2018 Sep 18;13(9):e0203702. doi: 10.1371/journal.pone.0203702. eCollection 2018. PMID 30226851
- [Derived] Cho DH, Joo HJ, Kim MN, Lim DS, Shim WJ, Park SM. Association between epicardial adipose tissue, high-sensitivity C-reactive protein and myocardial dysfunction in middle-aged men with suspected metabolic syndrome. Cardiovasc Diabetol. 2018 Jun 30;17(1):95. doi: 10.1186/s12933-018-0735-7. PMID 29960588
- [Derived] Joo HJ, Cho SA, Cho JY, Lee S, Park JH, Yu CW, Hong SJ, Lim DS. Different Relationship Between Physical Activity, Arterial Stiffness, and Metabolic Status in Obese Subjects. J Phys Act Health. 2017 Sep;14(9):716-725. doi: 10.1123/jpah.2016-0595. Epub 2017 May 17. PMID 28513244